CLINICAL TRIAL: NCT01561638
Title: Pulsed Radiofrequency Versus New Technique "Pulsed Dose" in Treatment of Chronic Shoulder Pain
Brief Title: Pulsed Radiofrequency Versus Pulsed Dose for Shoulder Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mohamed R El Tahan (Other)
Responsible Party: Sponsor-Investigator, Mohamed R El Tahan, Prof., Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anesth_MUH_6/2011
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Unilateral Chronic Shoulder Pain; Bilateral Chronic Shoulder Pain
Keywords: Pulsed; radiofrequency; single-dose; shoulder pain; Pain lasts more than one month; patients referred to the pain clinic from the shoulder clinic; Failed all conservative therapies available
MeSH Terms: conditions — Shoulder Pain | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group p (Active Comparator): pulse radiofrequency lesioning
  Interventions: Procedure: Conventional Radiofrequency
- sham group (Placebo Comparator): Controlled, conventional
  Interventions: Procedure: Sham
- group C (Active Comparator): Pulse dose radiofrequency
  Interventions: Procedure: Pulsed Dose Radiofrequency

INTERVENTIONS:
Procedure: Conventional Radiofrequency — pulsed radiofrequency will delivered at 45V for 2 cycles of 120 seconds(temperature not more than 42degree centigrade)
  Arms: group p
Procedure: Pulsed Dose Radiofrequency — pulsed dose pulsed radiofrequency,we will set the machine to give 480 pulses each pulse of 45 volts for 20 milliseconds duration with a temperature limit of 42 degree centigrade)
  Arms: group C
Procedure: Sham — will receive puncture for 4 minutes
  Arms: sham group

SUMMARY:
The "pulsed dose" RF treatment in various painful disorders may provides better pain relief with longer duration compared to previous Pulsed Radiofrequency (PRF) treatment in similar clinical settings. Also, there would has not been any worrisome complications from the procedures.

DETAILED DESCRIPTION:
Pain scores on visual analog scale (VAS) of 0_10 before and two hours immediately after radiofrequency lesioning and at 30 , 60, 90 day after procedure. Along with Oxford shoulder score (OSS) is a 12-item patient-reported specifically designed and developed for assessing outcomes of shoulder surgery e.g. for assessing the impact on patients' quality of life of degenerative conditions such as arthritis and rotator cuff problems. . The reduction in medications and the number of complications associated with the technique will be assessed.

Diagnostic suprascapular nerve block will done by 1.0 ml of 0.5% bupivacaine under fluoroscopic guidance using non-ionized dye (iohexol). Pain reduction more than 50% based on mean VAS assessment for at least three hours consider diagnostic.

Machine used is,(NeuroTherm 1100) RF lesion generator. The standard radiofrequency technique used, patient in sitting position , non-invasive blood pressure and peripheral oxygen saturation will monitored with non invasive pulse oxymetry. Vascular peripheral intravenous routes will opened shoulder region exposed and under complete aseptic technique skin will be anesthetized with 2.0 ml of 2% lidocaine at puncture site, suprascapular notch was identified. The landmark to guide the initial entry point was a line drawn along the length of the scapular spine, bisected with a vertical line from the angle of the scapula. A radiofrequency needle was introduced through the skin, 2.5 cm along the line of the spine in the upper outer quadrant, and then guided to the edge of the suprascapular notch by use of C_arm guide fluoroscopy with the image intensifier (22-gauge, 50-mm needle; 5-mm active tip) The nerve was located accurately by stimulating at 2 Hz (threshold < 0.5 V). PRF was applied for 120 seconds 2 or 3 times (NeuroTherm radiofrequency lesion generator) creating a tingling and paresthesia felt in the dermatomal distribution of the nerve in question. Motor stimulation (2 HZ). Impedances were checked to ensure a complete electrical circuit and range from 200 to 400 Ohms, if impedance is > 400 1 ml of 1% lidocaine will be injected.

ELIGIBILITY:
Inclusion Criteria:

* aged at least 18 years old
* both male and female
* had unilateral or bilateral chronic shoulder pain longer than one month
* rotator cuff tear arthropathy
* adhesive capsulitis shoulder instability
* post-traumatic pain
* post-surgical pain

Exclusion Criteria:

* Duration of shoulder pain < 1 month
* Patients had any previous surgical intervention or nerve blocks to the shoulder.
* patient refused or declined treatment
* Allergy to local anesthetics or steroid or contrast material.
* Severe psychiatric illness disorder,
* infection at site of injection
* Patients with a pacemaker or neurostimulator.
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pain | up to 3 months from the procedure
  reduction of pain immediately and one ,two, and three month .after procedure

SECONDARY OUTCOMES:
Side effects | up to12 weeks after the procedure
  Assessment of short term side effects and persisting side effects such as nausea, headache, momentary increase in pain, fever, tingling, itching, chest pain and/or burning skin at point of treatment
Shoulder Symptoms | up to12 weeks from the procedure
  Patient Self-Assessment of Shoulder Symptoms Before and After procedure Subjective symptoms would be recorded before procedure, and two hours after procedure, at four weeks, eight weeks, and twelve weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt